CLINICAL TRIAL: NCT03920540
Title: Phase 3, Double-blind, Randomized, Active-controlled (Part 1) and Open-labeled, Historical Placebo Controlled (Part 2) Study to Evaluate the Efficacy of Hunterase (Idursulfase-beta) in Hunter Syndrome (Mucopolysaccharidosis II) Patients
Brief Title: A Study of GC1111 in Hunter Syndrom Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GC1111_P3
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Hunter Syndrome
Keywords: GC1111; Mucopolysaccharidosis II; MPS II; idursulfase-beta; IDS
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC1111 (Experimental): In part 1, all participants who randomized into GC1111 arm should receive the GC1111 for 52 weeks.
  In part 2, all enrolled participants should receive the GC1111 for 52 weeks.
  Interventions: Combination Product: GC1111
- Comparator (Part 1) (Active Comparator): In Part 1, all participants who randomized into comparator arm should receive the GC1111 for 52 weeks.
  Interventions: Combination Product: Comparator

INTERVENTIONS:
Combination Product: GC1111 — GC1111 is 0.5mg per kg of body weight once weekly to be administered slowly by intravenous infusion.
  Arms: GC1111
Combination Product: Comparator — Comparator is 0.5mg per kg of body weight once weekly to be administered slowly by intravenous infusion.
  Arms: Comparator (Part 1)

SUMMARY:
The objective of this study is to evaluate the efficacy of GC1111 in Hunter Syndrome Patients

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Hunter syndrome
* Male at the age of ≥ 5
* Adequate abilities (including 6-MWT) to participate in this study in the opinion of the investigator.
* Voluntarily signed written informed consent to participation in this study
* Consent to contraception

Exclusion Criteria:

* Prior treatment with iduronate-2-sulfatase ERT
* History of bronchotomy, bone marrow trasplanation, or cord blood transplanation.
* Known hypersensitivity reactions to any of the components of the invetigational product
* Prior or planned administration of other investigational products within 30 days before treatment with the investigational product in this study or duirng this study.
* Unable to perform 6-MWT.
* Female

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Change in 6-MWT | at Week 53 from baseline

CONTACTS AND LOCATIONS:
Overall Officials: DongKyu Jin, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsug Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided